CLINICAL TRIAL: NCT03564028
Title: Effects of Energy Conservation Technique During Stair Climbing in COPD Patients : a Randomized Controlled Trial
Brief Title: Energy Conservation Technique in COPD Patients
Acronym: UpstAIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier du Havre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2018-A00566-49
Record Dates: First submitted 2018-06-11; First posted 2018-06-20 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; daily activity; stair climbing; rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Patients will perform two stair climbing sessions (each session include 108 steps) under two different conditions on the same day with at least 30 minutes of rest between the two sessions.
  the order of the two conditions will be randomly assigned
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- energy conservation technique (Experimental): Patients will perform one session of stair climbing of 108 steps (corresponding to 6 floors).
  Interventions: Other: energy conservation technique
- Control session (Other): Patients will perform one session of stair climbing of 108 steps (corresponding to 6 floors).
  Interventions: Other: control session

INTERVENTIONS:
Other: energy conservation technique — During the session of stair climbing, patients will perform a break at least of 5 seconds every 3 steps.
  Arms: energy conservation technique
Other: control session — Patients will realize one session of stair climbing at their own pace
  Arms: Control session

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is characterised by non-reversible bronchial obstruction associated with systemic disorders and comorbid factors. Dynamic hyperinflation during an exercise increase dyspnea and can reduce exercise capacity. Stair climbing is associated with prolonged dynamic hyperinflation and severe dyspnea in COPD patients. The aim of this study is to carry out the effect of an energy conservation technique on dyspnea to facilitate stair climbing.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of COPD
* Dyspnea in daily living (2-4 on the modified medical research council dyspnea scale)
* clinically stable

Exclusion Criteria:

* exercise contraindication Any musculoskeletal problems, cardiovascular or neurological comorbidities that limits exercise.
* exacerbation during the study
* inability to climb 6 floors

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-03-29 (Actual)

PRIMARY OUTCOMES:
Difference in Dyspnea at iso time and at time limit between the two sessions | The outcome will be measured before, at the end and every one minute during the stair climbing sessions. The two stair climbing sessions will perform the same day, separate from 30 minutes minimum for a total time frame of 1 day.
  Difference in dyspnea using Modified Borg Scale (0 - 10 points) 0=no dyspnea ; 10 = maximal effort

SECONDARY OUTCOMES:
difference in time required for the patient to climb the 6 floors | The outcome will be collected at the end of each sessions. The two stair climbing sessions will perform the same day, separate from 30 minutes minimum for a total time frame of 1 day.
  Difference in time (seconds) will be evaluated using a stopwatch
Difference in respiratory rate | Data will be continuously collected during every sessions. The two stair climbing sessions will perform the same day, separate from 30 minutes minimum for a total time frame of 1 day.
  Difference in respiratory rate (cycles per minute) will be measured breath-by-breath using a Respiratory Inductive Plethysmography
Difference in inspiratory capacity | The outcome will be collected before and at the end of each sessions (within 2 minutes after the end). The two stair climbing sessions will perform the same day, separate from 30 minutes minimum for a total time frame of 1 day.
  Difference in inspiratory capacity (Liters) will be measured using a portable spirometer
Difference in Cardiac Frequency | Data will be continuously collected during every sessions. The two stair climbing sessions will perform the same day, separate from 30 minutes minimum for a total time frame of 1 day.
  Difference in Cardiac Frequence (bpm) using a pulse oximetry
Difference in Oxygen Saturation | Data will be continuously collected during every sessions. The two stair climbing sessions will perform the same day, separate from 30 minutes minimum for a total time frame of 1 day.
  Difference in Oxygen Saturation
Difference in peripheral muscle oxygenation | Data will be continuously collected during every sessions. The two stair climbing sessions will perform the same day, separate from 30 minutes minimum for a total time frame of 1 day.
  Muscle oxygenation (arbitrary unit) will be evaluated using Near-infrared spectroscopy technology.
Difference in tidal volume | The outcome will be collected before and at the end of each sessions (within 2 minutes after the end). The two stair climbing sessions will perform the same day, separate from 30 minutes minimum for a total time frame of 1 day.
  Difference in tidal volume (Liters) will be measured breath-by-breath using a portable spirometer
Difference in muscular fatigue | The outcome will be measured before, at the end and every one minute during the stair climbing sessions. The two stair climbing sessions will perform the same day, separate from 30 minutes minimum for a total time frame of 1 day.
  Difference in muscular fatigue using Modified Borg Scale (0 - 10 points) 0=no muscular fatigue ; 10 = maximal effort

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier du Havre, Le Havre, Normandy, France

IPD SHARING:
Plan to Share IPD: Yes
Data will be available after publication. Please contact Guillaume Prieur at gprieur.kine@gmail.com

REFERENCES:
- [Derived] Prieur G, Combret Y, Medrinal C, Arnol N, Bonnevie T, Gravier FE, Quieffin J, Lamia B, Reychler G, Borel JC. Energy conservation technique improves dyspnoea when patients with severe COPD climb stairs: a randomised crossover study. Thorax. 2020 Jun;75(6):510-512. doi: 10.1136/thoraxjnl-2019-214295. Epub 2020 Mar 26. PMID 32217783